CLINICAL TRIAL: NCT06467292
Title: Sensorimotor Basis of Speech Motor Learning and Retention
Brief Title: Speech Motor Learning and Retention (Master Protocol)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000037622; 1R01DC022097-01A1 (NIH)
Record Dates: First submitted 2024-06-13; First posted 2024-06-21 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Speech
Keywords: Speech Motor Learning; Retention
MeSH Terms: conditions — Speech | interventions — Acclimatization; Transcranial Magnetic Stimulation; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Healthy right-handed adults with normal hearing will be recruited in equal number from both sexes. All participants will be fluent English speakers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Speech Motor Learning and Retention Aim 1 (Experimental): Aim 1: Participants will perform learning tasks while receiving altered/unaltered auditory feedback with cTBS applied to the appropriate area of the brain following learning. Retention of learning is assessed 24 hours later.
  Interventions: Device: continuous theta-burst stimulation (cTBS); Behavioral: Adaptation
- Speech Motor Learning and Retention Aim 2 (Experimental): Aim 2: Participants will perform learning tasks combined with shifted auditory feedback. Motor cortical excitability will be measured using single-pulse TMS to elicit motor evoked potentials.
  Interventions: Behavioral: Adaptation; Device: Single pulse Transcranial magnetic stimulation (TMS)
- Speech Motor Learning and Retention Aim 3 (Experimental): Aim 3: Participants will have fMRI with behavioral measures of speech motor learning.
  Interventions: Behavioral: Adaptation; Device: fMRI

INTERVENTIONS:
Device: continuous theta-burst stimulation (cTBS) — cTBS stimulation will be applied to different areas of the brain following learning. Stimulation will take place following learning in order to block motor memory retention.
  Arms: Speech Motor Learning and Retention Aim 1
Behavioral: Adaptation — Auditory adaptation in speech
Device: Single pulse Transcranial magnetic stimulation (TMS) — TMS will be delivered 10 times in each motor evoked potentials (MEP) recording block.
  Arms: Speech Motor Learning and Retention Aim 2
Device: fMRI — To assess functional connectivity patterns between regions that predict learning.
  Arms: Speech Motor Learning and Retention Aim 3

SUMMARY:
The overall goal of this research is to test a new model of speech motor learning, whose central hypothesis is that learning and retention are associated with plasticity not only in motor areas of the brain but in auditory and somatosensory regions as well.

DETAILED DESCRIPTION:
Aim 1 involves tests of speech motor memory retention following disruption of left hemisphere brain activity in either auditory, somatosensory or motor cortex or to a control site (hand area motor cortex right hemisphere). Continuous theta-burst stimulation (cTBS) is delivered following adaptation to altered auditory feedback to assess its effects on the retention of new learning.

Aim 2 assesses the temporal order in which plasticity occurs in cortical motor and sensory brain areas during speech motor learning.

In Aim 3, resting-state fMRI will be interleaved with speech motor adaptation. For information specific to each aim, please refer to the below corresponding, separate, clinicaltrials.gov records: unique IDs: 2000037622_a for Aim 1, 2000037622_b for Aim 2 and 2000037622_c for Aim 3.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Right-handed
* Normal hearing
* No speech disorder or reading disability

Exclusion Criteria:

* Cardiac pacemaker
* Aneurysm clip
* Heart or Vascular clip
* Prosthetic valve
* Metal implants
* Metal in brain, skull, or spinal cord
* Implanted neurostimulator
* Medication infusion device
* Cochlear implant or tinnitus (ringing in ears)
* Personal and/or family history of epilepsy or other neurological disorders or history of head concussion
* Psychoactive medications
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech motor learning | Performance as measured at the end of learning (30 minute session)
  Audapter software will be used to alter the first and second formant frequencies of the spoken words and this is played back to subjects through headphones. Subjects will be tested both with unaltered feedback and with abruptly introduced frequency shifts.The change in the first (F1) and second format frequency (F2) values will be assessed using Praat.
Retention of learning | 24 hours after learning (re-test lasts 30 minutes)
  The retention of adaptation to altered auditory feedback (and relearning) will be quantified in terms of F1 and F2 frequency shifts (relative to pre-training baseline). Larger values indicate more complete relearning or retention.

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No